CLINICAL TRIAL: NCT02219763
Title: A Longitudinal Study to Investigate the Effects of a 14-visit Comprehensive Lifestyle Weight Management Program on Body Weight and Quality of Life
Brief Title: The Effects of a Weight Management Program on Body Weight and Quality of Life
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Goedkoop, Sonja, Registered Dietitian, Massachusetts General Hospital
Other Study IDs: 2014P001032
Record Dates: First submitted 2014-08-15; First posted 2014-08-19 (Estimated); Last update posted 2014-08-19 (Estimated); Status verified 2014-06

CONDITIONS: Overweight; Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Evaluate the impact of a 12-week behavioral weight management program on body weight and quality of life. We hypothesize that participants will lose body weight and see improved quality of life after program completion.

DETAILED DESCRIPTION:
This study will evaluate weight change and quality of life among individuals after completion of a 12-week comprehensive group weight management program. Findings from this study will also help with program development and improvement within our center. The already established weight management program is called Healthy Habits for Life (HHL) and includes a total of 14 visits (one individual visit both before and after the 12 group sessions).

All patients who are enrolled in the Healthy Habits for Life group program at the Weight Center have an individual visit with a registered dietitian prior to beginning the group as part of standard care. At this visit the dietitian will obtain informed consent for participation in the research study and provide subjects consenting to participate in the study with the IWQOL-lite quality of life questionnaire.

After completion of the 12 HHL group sessions, all patients at the Weight Center have another individual visit with the dietitian to review weight and behavior changes since the initial evaluation. At this visit, subjects participating in the research study will again be provided with the IWQOL-lite questionnaire to fill out.

ELIGIBILITY:
Inclusion Criteria:

* English speaking adults aged 18 or older
* BMI ≥ 25
* Enrolled in HHL program at the MGH Weight Center

Exclusion Criteria:

* Non-English speaking patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (over age 18) with a BMI ≥ 25 enrolled in the 12-week Healthy Habits for Life (HHL) group program from the MGH Weight Center will be recruited. Subjects will be recruited over a 5-month period.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-06; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Weight Change | Approximately 4 months after enrollment
  The primary outcomes will be change in body weight comparing body weight at the start of the behavior change program and at the end. This includes weight at the initial individual visit, weights at each of the 12 group visits and body weight at the end of the group program.

SECONDARY OUTCOMES:
Quality of Life | Approximately 4 months after enrollment
  Quality of life will be assessed with a validated questionnaire at the start of the group and after completion of the group program.

OTHER OUTCOMES:
Blood laboratory values | Approximately 4 months after enrollment
  Labs collected include: Albumin, Alkaline Phosphatase, Total Bilirubin, Total Protein, ALT, AST, HbA1C, Lipids and Insulin. These labs will be collected at a patients first visit to the Weight Center and again after completion of the group program.

CONTACTS AND LOCATIONS:
Overall Officials: Sonja S Goedkoop, MSPH, RD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH Weight Center, Massachusetts General Hospital, Boston, Massachusetts, United States